CLINICAL TRIAL: NCT04150055
Title: Piloting an mHealth Mindfulness Therapy Intervention to Alleviate Symptoms of Stress for Caregivers of Older Adults With Cognitive Impairment.
Brief Title: mHealth Mindfulness for Dementia Caregivers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Principal Investigator, Elissa Kozlov, Ph.D, Core Faculty, Instructor, Rutgers, The State University of New Jersey
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro2019001438; KL2TR003018 (NIH)
Record Dates: First submitted 2019-10-30; First posted 2019-11-04 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-09

CONDITIONS: Caregiver Burnout; Stress; Anxiety
Keywords: mindfulness; caregiver; palliative care
MeSH Terms: conditions — Caregiver Burden; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Everyone in the study will get Mindfulness Coach and an orientation session. Mindfulness Coach is a self-guided mHealth intervention designed to help individuals learn MT, an evidence-based treatment to enhance health, wellness and mental health. The intervention will be introduced during 1 in-person session by a trained research assistant with 1-2 booster instructional phone call at 7 and 14-days to ensure that the participant knows how and is encouraged to use the app. The participant will also be provided with a laminated card that provides the basic instructions. We will encourage the participant to use Mindfulness Coach weekly for 8 weeks, or more if desired, as this treatment dose is commensurate with most in-person MT psychotherapy treatment protocols.
  Interventions: Behavioral: Mindfulness Coach

INTERVENTIONS:
Behavioral: Mindfulness Coach — Mindfulness Coach is an mHealth delivered mindfulness therapy.

SUMMARY:
The investigators will recruit 60 family caregivers of older adults with cognitive impairment or dementia to participate in a pilot feasibility and acceptability trial of Mindfulness Coach, an mHealth mobile application that delivers mindfulness therapy. Mindfulness Coach is a self-guided mHealth intervention designed to help individuals learn MT, an evidence-based treatment to enhance health, wellness and mental health. The app also offers a library of information about MT (e.g., "how to anchor participants' attention"), 12 audio-guided mindfulness exercises, and a catalog of additional exercises available for free. In addition to collecting data about the feasibility and acceptability of Mindfulness Coach with caregivers of patients with dementia or cognitive impairment, the investigators will also collect data on preliminary efficacy of Mindfulness Coach at relieving symptoms of caregiver burden, anxiety, stress and depression.

DETAILED DESCRIPTION:
The objective of this project is to evaluate the feasibility, acceptability and preliminary efficacy of Mindfulness Coach for stress and caregiver burden in caregivers of persons with dementia. The investigators will recruit participants across three outpatient geriatric primary care sites in the RWJ Barnabas Healthcare system: Monmouth, Monroe and New Brunswick.

Mindfulness Coach is a self-guided mHealth intervention designed to help individuals learn MT, an evidence-based treatment to enhance health, wellness and mental health. The app also offers a library of information about MT (e.g., "how to anchor your attention"), 12 audio-guided mindfulness exercises, and a catalog of additional exercises available for free. The app tracks progress over time with a mindfulness mastery assessment, has customizable reminders which the patient will learn to set during orientation, and goal-setting and tracking features, which the patient will learn to customize during orientation. Mindfulness Coach was designed by a multidisciplinary team of experts in telehealth, technology and mental health from the VA's National Center for PTSD and the Department of Defense's National Center for Telehealth and Technology and is free and available on iOS and Android. In this study, the intervention will be introduced during 1 in-person session by a trained research assistant with 1-2 booster instructional phone call at 7 and 14-days to ensure that the participant knows how and is encouraged to use the app. The participant will also be provided with a laminated card that provides the basic instructions. The investigators will encourage the participant to use Mindfulness Coach weekly for 8 weeks, or more if desired, as this treatment dose is commensurate with most in-person MT psychotherapy treatment protocols.

Subjects and Sample Size:The investigators will recruit 60 patients from three RWJ Barnabas sites: Monmouth, Monroe and New Brunswick. Caregivers will be recruited by physician referral. Physicians will identify patients with a diagnosis of dementia or cognitive impairment and their family caregivers. The term "family caregiver" refers to any family member or relative who is involved in a patient's health care because of a personal connection, not for financial compensation. Family caregivers are eligible if they are age 21 or older, English-speaking, currently own a mobile device (smartphone or tablet) and spend at least 10 hours per week providing care to the older adult patient. Procedures: Providers will notify study coordinator of patients who have a diagnosis of dementia or cognitive impairment and typically have a family caregiver present during medical visits. Emails will be sent to providers to inquire about potential subjects. The study research assistant (RA) will call potential subjects to obtain consent for a phone screen. The screen will include questions about current caregiving practices and questions about mobile device usage (e.g., do participants own a smart phone or tablet? How often do participants use this device?). If a patient is eligible and interested in participating, an in-person baseline assessment and orientation will be scheduled at the primary care provider's office. Informed consent will be obtained in person prior to the baseline assessment. The baseline assessor will also be the individual who orients participants to Mindfulness Coach. Follow-up interviews will be conducted via telephone.

The orientation will consist of the following components: 1.) education about the app, its developers and MT (to establish credibility); 2.) discussion of goals of the app; 3.) procedural information about how to launch and navigate the app; and 4.) assessment of participant's ability to use the app: participants must be able to meet pre-established criteria of being able to open, launch, navigate and use the app independently prior to the end of the orientation session. During orientation, study personnel will discuss the benefits of daily, brief (5-15 minutes) mindfulness practice and ask participants if daily practice is a goal they would be willing to set. If the participant is amenable, study personnel will help participants set reminders (push notifications) within Mindfulness Coach to facilitate daily practice. The investigators will work with each participant to set mindfulness practice goals that are tailored to the unique needs of each participant. Participants will also be given a laminated instructional card explaining how to access and use Mindfulness Coach. Booster sessions: The study RA will schedule a 1-week booster phone call with intervention participants to troubleshoot potential difficulties users may be experiencing with the application. At this session, participants will be asked if they have used the app in their first week. If they have not, the investigators will schedule an additional follow up booster session phone call at 2-weeks to provide additional troubleshooting and encouragement.

ELIGIBILITY:
Inclusion Criteria:

* owns a smart phone or tablet
* speaks English fluently, aged 21+
* identifies as the caregiver for an older adult with dementia or mild cognitive impairment

Exclusion Criteria:

* does not own smart phone or tablet
* does not speak English fluently
* is under age 21
* does not provide care for older adult with dementia or mild cognitive impairment.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-11-05 (Actual); Primary Completion 2021-03-08 (Actual); Study Completion 2021-03-08 (Actual)

PRIMARY OUTCOMES:
Feasibility - amount of time participants spend in app | 8 weeks
  how much do caregivers use mindfulness coach
Acceptability - satisfaction with mindfulness coach survey | 8 weeks
  Do caregivers find mindfulness coach helpful and easy to use?
Bakas Caregiver Outcomes Scale - 15 items | 8 weeks
  scores range from 15-105 with higher scores indicating better outcomes

SECONDARY OUTCOMES:
hospital anxiety and depression scale- anxiety sub scale | 8 weeks
  scores range from 0-21 with higher scores indicating worse outcomes
hospital anxiety and depression scale, depression sub scale | 8 weeks
  scores range from 0-21 with higher scores indicating worse outcomes
The World Health Organization Quality of Life Brief | 8 weeks
  scores range from 26-130 with higher scores indicating better outcomes
perceived stress scale | 8 weeks
  scores range from 0-40 with higher scores indicating worse stress

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - RWJ Barnabas Monmouth South, Lakewood, New Jersey
  - RWJ Barnabas, Monroe, New Jersey

IPD SHARING:
Plan to Share IPD: No